CLINICAL TRIAL: NCT01887756
Title: Research and Clinical Aspects of the Project Study of Home Based Tele-Rehabilitation Program for Patients With Stroke
Brief Title: Research Online Tele-Rehabilitation Program in People After a Stroke Living at Home
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Halted before intervention due to approval of service.
Sponsor: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Dr. Shlomo Flechter, Principal Investigator, Clalit Health Services
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTR-Motion
Record Dates: First submitted 2013-06-12; First posted 2013-06-27 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2013-06

CONDITIONS: Stroke
Keywords: telerehabilitation stroke virtual reatlity
MeSH Terms: conditions — Stroke | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm study (Experimental): The clients will receive tele-rehabilitation treatment via the Gertner Tele-Motion Rehabilitation system with remote online monitoring by the therapist. Treatment feedback is given in the form of Knowledge of results (game scores) and Knowledge of performance (feedback of compensatory movements made while using the upper extremity) to enhance motor learning. The software generates a report which includes the duration and type of exercises performed by the subject.
  Interventions: Device: Tele Rehabilitation

INTERVENTIONS:
Device: Tele Rehabilitation
  Other Names: Gertner Institute Tele Motion Rehabilitation system

SUMMARY:
Telerehabilitation refers to the use of Information and Communication Technologies (ICT) to provide rehabilitation services to people remotely in their homes or other environments. By using ICT, patient access to care can be improved and the reach of clinicians can extend beyond the physical walls of a traditional healthcare facility, thus expanding continuity of care to persons with disabling conditions. The concept of telecare, when telerehabilitation is used to deliver services to patients in their homes or other living environments, empowers and enables individuals to take control of the management of their medical needs and interventions by enabling personalized care, choice and personal control Research Goal and Objectives

1. To investigate the clinical feasibility and usability of the Gertner Tele-Motion-Rehab system in post-stroke patients, in their homes.
2. To evaluate Gertner Tele-Motion-Rehab system clinical improvement within the patient's home in terms of:

   1. function of the weak upper extremity
   2. performance of ADL

ELIGIBILITY:
Inclusion Criteria:

* 6-72 months post stroke
* Sitting balance intact (ability to go beyond the midline of the body)
* Moderate impairment of the affected upper extremity determined by range of motion (ROM); shoulder flexion and abduction must be more than 45 degrees with mild to moderate compensations; elbow flexion should be about 45 degrees and trunk movement of about 10 cm.
* Basic ability to independently use the tele-system via touching virtual objects on the screen.
* Having a personal computer (at least Intel i3 processor, with Win7 operating system),Internet access (10MBps) and a large computer monitor (at least 26") at home.
* Caregiver, available when needed, toprovide support throughout the intervention.

Exclusion Criteria:

* Other medical conditions limiting participation in low-intensity exercise training.
* Major receptive aphasia and screening criteria consistent with dementia (Mini-MentalState score <24).
* Untreated major depression.
* Presence of unilateral spatial neglect as determined by star cancellation (score less than 51).
* Hemianopsia
* Apraxia (limb and ideomotor)
* Other medical conditions that affect the central or peripheral nervous system
* Ataxia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
System usability scale | Second assessment (after 6 weeks)
  This questionnaire includes 10 items which provide a global view of subjective assessment of a system's usability. Each item was rated on a five-point scale from one (disagree totally) to five (agree totally). Five items are positive statements, such as "I think that I would like to use this system frequently" and "I thought the system was easy to use" and the other five items are negative, for example, "I found the system unnecessarily complex" and "I think that I would need the support of a technical person to be able to use this system." The item scores were calculated to give an overall score ranging from 10 to 100 points. The SUS has been shown by the authors to be a robust and reliable evaluation tool but its psychometric properties have not been fully investigated. (Brooke et al., 1995)
Short Feedback Questionnaire | Second assessment ( after 6 week)
  This is an 8-item questionnaire which queries the user's sense of presence, perceived difficulty of the task and any discomfort that users may have felt during the experience. The first six items assess the participant's (1) feeling of enjoyment, (2) sense of being in the environment, (3) success, (4) control, (5) perception of the environment as being realistic and (6) whether the feedback from the computer was understandable. The seventh item queries whether participants felt any discomfort during the experience. An eighth item queries their perceived difficulty while performing the task. Responses to the first seven items are rated on a scale of 1-5 where 1=not at all and 5 = very much. Responses to the eighth item is also rated on a 1-5 scale where 1= very easy and 5= very difficult. A total mean score for each participant will be calculated for the first six items.(Kizony et al., 2006)
Fugl-Meyer Assessment upper extremity part (FMA) | First assessment (beginning)
  The FMA assesses the motor impairment of the upper extremity after stroke. Each movement is graded on a 3-point scale, and the total score for the upper extremity ranges from 0-60 points where a higher score represents more active movements. An additional part assesses the coordination of the affected upper extremity and the score ranges between 0-6 where a higher score represents poorer coordination ability. This test is one of the most commonly used instruments in rehabilitation and its validity and reliability have been well established (Fugl-Meyer et al., 1975; Wood-Dauphinee, Williams, & Shapiro, 1990; Chae, Johnston, Kim, &Zorowitz, 1995).
Motor Activity Log | First assessment (beginning)
  The Mal consist of a semi structured interview for the patient to assess the use of the paretic arm and hand during activities of daily living. Two scores are given for each activity, 1 for the amount of use (AOU) and 1 for the quality of movement (QOM). The questions concern activities performed during the past week or, occasionally, the past year. Possible scores range from 0 (never use the affected arm for this activity) to 5 (always use the affected arm for this activity). (Van der Lee, Beckerman, Knol, de Vet, Bouter, 2004)
Change in System Usability Scale between 6th week and 12th week | Third assessment (after 12 weeks)
Change in Short Feedback Questionnaire between 6th week and 12th week | Third assessment (after 12 weeks)
Change in Fugl-Meyer Assessment upper extremity part (FMA)between baseline and 6th week | Second assessment (after 6 weeks)
Change in Fugl-Meyer Assessment upper extremity part (FMA)between 6th week and 12th week | Third Assessment (after 12 weeks)
Change in Motor Activity Log between baseline and 6th week | Second assessment (after 6 weeks)
Change in Motor Activity Log between 6th week and 12th week | Third assessment (after 12 weeks)

SECONDARY OUTCOMES:
Range of Motion (ROM) of shoulder and elbow | First, second and third assessments (beginning, 6 & 12 weeks respectively)
  Standard clinical goniometer will be used to measure changes in shoulder (abduction and flexion) and elbow flexion Range of Motion angles in degrees.
Visual Analog Scale (VAS) | Second and third assessments (6 & 12 weeks respectively)
  for Pain evaluation will be used to document pain intensity, and rated from 0 to 10. The VAS is a 10 cm line representing pain intensity from "no pain" (0) to "worst pain" (10). Subjects will be requested to bisect the line at the point that best represented their level of neck pain. The VAS has been recognized as a generic pain intensity instrument for over two decades (Langley & Sheppard, 1985) and has been found valid and sensitive to changes in acute (Breivik et al., 2000) and chronic (Ogon et al., 1996) pain.
Instrumental Activities of Daily Living (IADL) | First and third assessments (beginning & 12 weeks respectively)
  A questionnaire which evaluates the subject's capacity to perform eight different IADL tasks such as cooking, the use of transportation, shopping and taking medication (Lawton & Brody, 1969; Lawton et al., 1982).
Functional Independence Measure (FIM) | First and third assessments (beginning & 12 weeks respectively)
  FIM rates the degree of disability and outcome after rehabilitation. It assesses 18 components of basic activities of daily living (e.g. dressing) and used here to characterize functional status. Thirteen activities (in areas of eating, dressing, grooming, bathing, toileting, transfers and mobility) constitute the motor part of the FIM and five (in areas of comprehension, expression, social relations, problem solving and memory) constitute the cognitive part of the FIM. Each activity is graded on a seven point scale with a total score range between 13-91 for the motor part and 5-35 for the cognitive part. The reliability and validity is well established (Granger, 1998). It was found suitable to use with patients who had a stroke (Ring et al., 1997; Granger Cotter, Hamilton & Fiedler, 1993) and also has been used for people with SCI (Sipski, Jackson, Gomez-Marin, Estores&Stein, 2004). (Hamilton Granger, Sherwin, Zielezny&Tashman, 1987).
Stroke Impact Scale (SIS) | First and third assessments (beginning & 12 weeks respectively)
  SIS is a self-report that each participant will complete regarding his or her overall quality of life, including perceived difficulties with activities of daily living (ADL). (University of Kansas, 2008, http://www2.kumc.edu/coa/ SIS/SIS_pg2.htm )

OTHER OUTCOMES:
NIHSS | Beginning
  The National Institutes of Health Stroke Scale (NIHSS) is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. the scale is widely used as a clinical assessment tool to evaluate acuity of stroke patients, determine appropriate treatment, and predict patient outcome. The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items. The single patient assessment requires less than 10 minutes to complete. (http://www.nihstrokescale.org/)
Behavioral Assessment of the Dysexecutive Syndrome (BADS) | Beginning
  This is a valid and reliable test battery aimed at predicting everyday problems arising from the dysexecutive syndrome (Norris & Tate, 2000). The Battery consists of 6 subtests which measures different aspects of executive functions; temporal judgment, rule shift cards, action program, key search, zoo map and modified six elements test (see appendix 5). For each subtest a profile score between 0 and 4 is calculated and all the scores are combined to a total profile score which is converted to an age-matched score. In addition the battery consists of a questionnaire; the Dysexecutive Functional Questionnaire (DEX) that assess how the deficits in executive functions manifest in everyday activities. This questionnaire is administered to the person who had a stroke as well as to his or her caregiver. (Wilson et al., 1996)

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Flechter, MD, Principal Investigator — Clalit Health Services
Locations (1):
- Neurology Department, Bat Yamon Medical Center, Bat Yam, Israel